CLINICAL TRIAL: NCT03099980
Title: Open-label, Investigator-Initiated, Single Site Exploratory Trial Evaluating Cosentyx (Secukinumab) for Patients With Moderate-to-Severe Hidradenitis Suppurativa
Brief Title: Exploratory Trial Evaluating Cosentyx (Secukinumab) for Patients With Moderate-to-Severe Hidradenitis Suppurativa
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAIN457AUS03T
Record Dates: First submitted 2017-03-29; First posted 2017-04-04 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-05

CONDITIONS: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — secukinumab

STUDY DESIGN:
Intervention Model Description: secukinumab 300 mg (2 x 150 mg pre-filled syringe) administered at Baseline, Weeks 1, 2, 3, 4, and then Q4W for 24 weeks via subcutaneous injections
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Secukinumab (Experimental): All participants will be assigned to receive secukinumab 300 mg (2 x 150 mg PFS subcutaneous injections) administered at Baseline, Weeks 1, 2, 3, 4, and then Q4W for 24 more weeks.
  Interventions: Biological: secukinumab

INTERVENTIONS:
Biological: secukinumab — secukinumab 300 mg (2 x 150 mg pre-filled syringe) administered at Baseline, Weeks 1, 2, 3, 4, and then Q4W for 24 weeks via subcutaneous injections
  Other Names: Cosentyx

SUMMARY:
This is a pilot study in which the the safety and feasibility of secukinumab in HS patients as well as information about the effect size will be determined in order to inform a future larger randomized control trial with an active comparator.

DETAILED DESCRIPTION:
Secukinumab is an antibody that inhibits Interleukin-17A, and IL-17 promotes neutrophil activities. Neutrophils are found in large numbers in HS. The expression of the inflammatory cytokines IL-17, IL-1β, and TNF-α were enhanced in lesional skin of HS patients.

Prior studies have demonstrated improvement in HS with biologic medications such as the tumor necrosis factor inhibitors adalimumab and infliximab. Studies have shown conflicting data regarding the efficacy of etanercept for HS and success with anakinra.

This is an initial pilot study of secukinumab for the purpose of studying how it may alter HS disease symptoms. This study is not intended to alter indications for drug use but may inform the design of an efficacy study that may alter FDA labeling changes in the future. There are limitations of this study that arise from it being a single-arm clinical trial with a small number of subjects. These limitations include the limited generalizability knowledge of this study due to the lack of an active comparator. However, the data obtained from this study will potentially be used to support the design of larger future randomized placebo controlled studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients must give written informed consent before any assessment is performed.
* Subject has moderate-to-severe HS as defined by: 1. HS lesions in at least 2 distinct anatomic areas, one of which is Hurley stage II or III on evaluation at Screening. 2. Stable HS for at least 2 months (60 days) prior to Screening and also at the Baseline visit as determined by the investigator.
* Total abscess and inflammatory nodule (AN) count of greater than or equal to 3 at the Baseline visit.
* Subject has had HS diagnosis for at least 3 months prior to Baseline.
* Subject must have failed at least one prior course of oral antibiotics.
* Subject must agree to daily use (and throughout the entirety of the study) of one of the following over-the-counter topical antiseptics on their body areas affected with HS lesions: chlorhexidine gluconate, triclosan, benzoyl peroxide, or dilute bleach in bathwater.
* Subject must be at least 18 years of age at time of Screening

Exclusion Criteria:

* Subject has had history of malignancy within the past 5 years
* Women who are pregnant, nursing, or planning pregnancy within 6 months after last subcutaneous injection. Male patients who are planning for their partner's pregnancies within 6 months from the last subcutaneous injection
* Subject has history of active TB. Subjects with latent TB must have been on treatment for at least 8 weeks prior to Baseline visit and the course of prophylaxis is planned to be completed.
* Subject has had infections requiring oral or intravenous (IV) antibiotics within 14 days prior to Baseline.
* Subject has significant serious medical problems or a condition that significantly immunocompromises the subject.
* Subject has had clinically significant hematological abnormalities defined as HGB <13.5 g/dL (<135 g/L) or a HCT <41.0 percent in men, or a value <12.0 g/dL (<120 g/L) or <36.0 percent in women.
* Subject has previously used secukinumab.
* Subject has had any other active skin disease or condition that may interfere with HS assessment.
* Subject has received prescription topical therapies for treatment of HS within 7 days prior to Baseline.
* Subject has received systemic non-biologic therapies with potential therapeutic impact for HS <14 days prior to Baseline visit.
* Clinically significant abnormal laboratory values as evaluated by the investigator.
* Patients with Crohn's disease or Ulcerative Colitis.
* Subject has received any systemic immunosuppressive treatment within 1 month prior to Baseline visit. Subject has received anti-TNF therapy within 3 months prior to Baseline visit. Subject has received anti IL-23 therapy within 3 months prior to Baseline visit.
* Subject has received intralesional steroid injection within 2 weeks prior to Baseline visit.
* Subject with known Human Immunodeficiency Virus (HIV) positive status or with positive HIV testing at Screening.
* Subjects with Hepatitis B and Hepatitis C positive status or with positive Hepatitis B and Hepatitis C testing at screening.
* Subjects with active cardiovascular disease or relevant risk factors such as prior myocardial infection or stroke.
* Subjects with chronic infection or a history of recurrent infections.
* Subjects with a history of latex allergy or sensitivity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-07-11 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Hidradenitis Suppurativa Clinical Response (HiSCR) | week 24
  percent of patients achieving clinical response

CONTACTS AND LOCATIONS:
Overall Officials: David Rosmarin, MD, Principal Investigator — Tufts Medical Center, Department of Dermatology
Locations (1):
- Tufts Medical Center, Department of Dermatology, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No